CLINICAL TRIAL: NCT03210987
Title: Effect of Bedside Patient Case Presentation Compared to Outside the Room Case Presentation on Patient Perception of Quality of Care and Patient Outcomes: a Randomized-controlled, Multicenter Trial
Brief Title: Effects of Bedside Compared to Outside the Room Case Presentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Aarau (Other); Kantonsspital Liestal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Visitenstudie (2017-00991)
Record Dates: First submitted 2017-06-27; First posted 2017-07-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Bedside Patient Case Presentation; Outside-the-room Patient Case Presentation
Keywords: ward round; patient case presentation; communication; patient-centered care
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: On the day before the ward round, patients will be randomized 1:1 into one of both study arms. In one study arm, patient case presentation will be performed at bedside. In the other study arm, patient case presentation will be performed outside the room.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient case presentation Bedside (Active Comparator): In the bedside presentation group, patient case presentation and discussions will be at bedside with direct involvement of the patient as needed.
  Interventions: Procedure: patient case presentation bedside
- patient case presentation Outside-the-room (Active Comparator): In the outside the room condition, case presentation and discussions will take place outside without the patient being present. After the case presentation and discussions the team will enter the room and give the patient a short summary of the medical situation, complete the medical information and examine the patient, as needed, and discuss the next steps.
  Interventions: Procedure: patient case presentation Outside-the-room

INTERVENTIONS:
Procedure: patient case presentation bedside — Patient case presentation in absence or presence of Patient at bedside.
  Other Names: teaching round; bedside round; ward round
  Arms: patient case presentation Bedside
Procedure: patient case presentation Outside-the-room — Patient case presentation Outside-the-room.
  Arms: patient case presentation Outside-the-room

SUMMARY:
Patient case presentations during ward rounds can take place at the bedside or outside the room. The best approach to patient case presentation is yet unclear. Thus, the overall aim of this multicenter, randomized-controlled study is to test the hypothesis that outside the room patient case presentation compared to bedside patient case presentation results in better outcomes across different dimensions including patient understanding and perception of quality of care as well as patient outcomes, physicians' preferences, perception of quality and effectiveness, and timing of the ward rounds, respectively.

DETAILED DESCRIPTION:
Patient-centered care may be defined as "providing care that is respectful of and responsive to individual patient preferences, needs, and values and ensuring that patient values guide all clinical decisions". Involving patients in all steps of the healthcare process is thus important. Yet, best presentation of patients' cases during ward rounds remains unknown. During outside the room patient case presentation, the medical team discusses difficult patient or medical issues in the team, and later presents a "patient-friendly" synthesis to the patient. Bedside patient case presentation, on the other hand, allows a patient to be part of the whole team discussion. Yet, there is concern that patients may be unable to cope with the magnitude of medical information and misunderstandings may occur. Currently, there is equipoise regarding both possibilities of patient case presentation with an important lack of trial data. We thus aim to compare the effect of bedside patient case presentation with outside the room patient case presentation during ward rounds ("Chefarztvisite") on different patient- and physician-related endpoints.

Therefore, this randomized controlled trial aims to test the hypothesis that outside the room patient case presentation compared to bedside patient case presentation results in better outcomes across different dimensions including patient understanding and perception of quality of care as well as patient outcomes, physicians' preferences, perception of quality and effectiveness, and timing of the ward rounds, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult (>18 years) medical inpatients during their first ward round independently of their underlying disease and reason for hospital stay.

Exclusion Criteria:

1. Patients with cognitive impairment, such as dementia/delirium
2. Patients with paracusia.
3. Patients who do not understand local language(s).
4. Patients already included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1092 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Subjective understanding of disease and management | post ward round up to 36 h
  average of the visual analog scale (VAS) score across the following three dimensions rated by the patient (0 "I have no knowledge at all about the situation" to 100 "I have best possible knowledge about the situation": I. Patients' subjective understanding of the disease II. Patients' subjective understanding of the therapeutic concept III. Patients' subjective understanding of the next steps

SECONDARY OUTCOMES:
Improvement understanding | post ward round up to 36 h
  Patients' perception about how well the current ward round improved the understanding of each of these three components, i.e., current disease, therapeutic concept, and next steps (VAS, 0-100)
Objective understanding of disease and management | post ward round up to 36 h
  Comparison of patients' recall information regarding current main diagnosis, main therapeutic measures and next steps (qualitative information) with medical chart information.
  Answers regarding current main diagnosis will be categorized as: (1) patient correctly states both pathophysiology and localization, (2) patient correctly states either pathophysiology or localization, (3) patient states neither pathophysiology nor localization (correctly) but correctly states symptoms, (4) patient correctly states that the current diagnosis is still unclear, (5) patient states incorrect information, (6) patient correctly states a secondary diagnosis relevant for the current hospitalization Answers regarding main therapeutic measures and next steps will be categorized as: (1) correct (regarding main diagnosis), (2) incorrect (regarding main diagnosis), (3) correct (regarding secondary diagnosis), (4) incorrect (regarding secondary diagnosis)
Overall quality of care | post ward round up to 36 h
  Patients' perception (each rated on a VAS 0-100) regarding: comprehensibility of information during ward round, satisfaction with care, confidence in the medical team, perceived competence of the medical team, perceived interpersonal behavior during ward round, affective response of the patients, adequacy of ward round duration (includes two additional questions asking for patients' estimations on how much time the medical team spent on their case within the ward round as well as on average per day (estimates in minutes))
Follow up health status | 30 days follow up after study inclusion
  Patients' perceived health status (EuroQol five dimensions questionnaire)
Follow up understanding | 30 days follow up after study inclusion
  Patients' subjective (VAS 0-100) and objective (recall as compared to objective medical chart information) understanding
Follow up quality of hospital care | 30 days follow up after study inclusion
  Patients' overall perspective of hospital care (Hospital Consumer Assessment of Healthcare Providers and Systems, HCAHPS)
Follow up readmission | 30 days follow up after study inclusion
  Patients' readmission rate since study inclusion
Follow up duration of hospitalization | 30 days follow up after study inclusion
  total duration of hospitalization
Treating team satisfaction | post ward round up to 96 h
  The treating team's satisfaction with ward round (rated on a VAS 0-100)
Treating team performance | post ward round up to 96 h
  The treating team's perceived performance in the ward round (each rated on a VAS 0-100): time management of the ward round, interaction within the medical team and with the patient during ward round, perceived time management and feasibility
Treating team affect | post ward round up to 96 h
  The treating team's affective response (rated on a VAS 0-100)
Treating team preference | post ward round up to 96 h
  The treating team's preference of bedside compared to outside the room patient case presentation (rated on a semantic differential ranging from 1 "I prefer bedside ward rounds" to 6 "I prefer ward rounds outside the room")
Timeliness | during ward round which may last from 5 up to 30 minutes
  duration of the ward round (minutes)
Communication-specific items during ward rounds | during ward round which may last from 5 up to 30 minutes
  Rated by investigator (nominal 3-point scale (1 = yes; 2 = no; 3 = not applicable): structuring of conversation, use of patient-centered techniques, use of physician-centered techniques, dealing with emotions, conveying of complex information, negotiation of shared concepts of disease and treatment, realization of shared decision making, breaking bad news

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hunziker, Prof., Principal Investigator — Medical Communication, Department of Psychosomatic Medicine, University Hospital Basel, and University of Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehmann LS, Brancati FL, Chen MC, Roter D, Dobs AS. The effect of bedside case presentations on patients' perceptions of their medical care. N Engl J Med. 1997 Apr 17;336(16):1150-5. doi: 10.1056/NEJM199704173361606. PMID 9099660
- [Background] Chauke HL, Pattinson RC. Ward rounds -- bedside or conference room? S Afr Med J. 2006 May;96(5):398-400. No abstract available. PMID 16751910
- [Background] O'Leary KJ, Killarney A, Hansen LO, Jones S, Malladi M, Marks K, M Shah H. Effect of patient-centred bedside rounds on hospitalised patients' decision control, activation and satisfaction with care. BMJ Qual Saf. 2016 Dec;25(12):921-928. doi: 10.1136/bmjqs-2015-004561. Epub 2015 Dec 1. PMID 26628552
- [Background] Ramirez J, Singh J, Williams AA. Patient Satisfaction with Bedside Teaching Rounds Compared with Nonbedside Rounds. South Med J. 2016 Feb;109(2):112-5. doi: 10.14423/SMJ.0000000000000419. PMID 26840968
- [Background] Seo M, Tamura K, Morioka E, Shijo H. Impact of medical round on patients' and residents' perceptions at a university hospital in Japan. Med Educ. 2000 May;34(5):409-11. doi: 10.1046/j.1365-2923.2000.00516.x. No abstract available. PMID 10760128
- [Derived] Gross S, Becker C, Beck K, Memma V, Gaab J, Schutz P, Leuppi JD, Schaefert R, Langewitz W, Trendelenburg M, Breidthardt T, Eckstein J, Osthoff M, Bassetti S, Hunziker S. Occurrence of sensitive topics during ward round: an ancillary analysis of the BEDSIDE-OUTSIDE trial. BMJ Open. 2023 Sep 21;13(9):e073584. doi: 10.1136/bmjopen-2023-073584. PMID 37734895
- [Derived] Becker C, Gross S, Gamp M, Beck K, Amacher SA, Mueller J, Bohren C, Blatter R, Schaefert R, Schuetz P, Leuppi J, Bassetti S, Hunziker S. Patients' Preference for Participation in Medical Decision-Making: Secondary Analysis of the BEDSIDE-OUTSIDE Trial. J Gen Intern Med. 2023 Apr;38(5):1180-1189. doi: 10.1007/s11606-022-07775-z. Epub 2022 Sep 9. PMID 36085211
- [Derived] Gross S, Beck K, Becker C, Gamp M, Mueller J, Loretz N, Amacher SA, Bohren C, Gaab J, Schuetz P, Mueller B, Fux CA, Leuppi JD, Schaefert R, Langewitz W, Trendelenburg M, Breidthardt T, Eckstein J, Osthoff M, Bassetti S, Hunziker S. Perception of physicians and nursing staff members regarding outside versus bedside ward rounds: ancillary analysis of the randomised BEDSIDE-OUTSIDE trial. Swiss Med Wkly. 2022 Jan 19;152:w30112. doi: 10.4414/smw.2022.w30112. eCollection 2022 Jan 17. PMID 35072414
- [Derived] Becker C, Gamp M, Schuetz P, Beck K, Vincent A, Hochstrasser S, Metzger K, Widmer M, Thommen E, Mueller B, Fux CA, Leuppi JD, Schaefert R, Langewitz W, Trendelenburg M, Breidthardt T, Eckstein J, Osthoff M, Bassetti S, Hunziker S; BEDSIDE-OUTSIDE Study Group. Effect of Bedside Compared With Outside the Room Patient Case Presentation on Patients' Knowledge About Their Medical Care : A Randomized, Controlled, Multicenter Trial. Ann Intern Med. 2021 Sep;174(9):1282-1292. doi: 10.7326/M21-0909. Epub 2021 Jun 29. PMID 34181449